CLINICAL TRIAL: NCT00457379
Title: Randomized, Clinical Trial to Study the Effect of Exercise Training on the Function of HDL-Cholesterol, Endothelial Function, Oxidative Stress and Regenerative Capacity of Endothelial Progenitor Cells in Patients With Coronary Artery Disease
Brief Title: Effect of Exercise Training on the Function of HDL-Cholesterol, Endothelial Function and Endothelial Progenitor Cells in Patients With Coronary Artery Disease (HERCET-Study)
Acronym: HERCET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 4031214
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; HDL-Cholesterol; Endothelial Function; Endothelial Progenitor Cells; normal blood HDL-Cholesterol level
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

INTERVENTIONS:
Behavioral: physical exercise

SUMMARY:
Patients with coronary artery disease are characterized by an increased cardiovascular risk and they often have low blood high density lipoprotein (HDL)-cholesterol levels or HDL-cholesterol with modified vasculoprotective properties.

The purpose of the present study is to characterize the quality of HDL-cholesterol in patients with coronary artery disease and normal blood HDL-cholesterol levels and to examine the effect of exercise training on the vasculoprotective effects of HDL-cholesterol in these patients. Additionally, the researchers aim to investigate the endothelial function, oxidative stress and the regenerative capacity of the endothelial progenitor cells in patients with coronary artery disease and the changes dependent on physical activity of patients.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease
* Normal HDL-cholesterol levels in blood:

  * > 40 mg/dl (1.03 mmol/L) in males
  * > 50 mg/dl (1.29 mmol/L) in females

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Acute coronary syndrome
* Unstable angina pectoris
* Myocardial infarction during the last 8 weeks
* Therapy with niacin
* Active infections
* Ventricular arrhythmias
* Systolic blood pressure > 160 mmHg or diastolic blood pressure > 95 mmHg
* Cancer
* Pregnant or lactating
* Alcoholism

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
vasculoprotective and regenerative functions of HDL-cholesterol before and after 8-weeks of exercise training

SECONDARY OUTCOMES:
flow-mediated, endothelium-dependent vasodilation of radial artery measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Drexler, MD, Study Director — Hannover Medical School; Ulf Landmesser, MD, Principal Investigator — Hannover Medical School; Kristina Sonnenschein, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany